CLINICAL TRIAL: NCT05227807
Title: The Efficacy of Mouth Exercise for Preventing Trismus in Oral Cancer Patients After Receiving Surgery and Radio or Chemotherapy
Brief Title: The Efficacy of Mouth Exercise in Oral Cancer Patients After Receiving Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Chang Gung Medical Foundation (Other)
Responsible Party: Principal Investigator, Tsae Jyy, Wang, professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 100-4007A3
Record Dates: First submitted 2021-12-12; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Neoplasms
Keywords: oral cancer; Trismus; Mouth-opening training; Maximum interincisal opening; Follow-up telephone calls; Mandibular function
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms; Trismus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): the control group received routine care.
  Interventions: Behavioral: Usual care
- Intervention group (Experimental): Intervention develop from the theoretical framework of social cognition theory
  Interventions: Behavioral: mouth opening exercise

INTERVENTIONS:
Behavioral: mouth opening exercise — The intervention group receives an oral exercise intervention, including a 30-minute individual training, a multimedia oral exercise education video along with a print education booklet, and three follow-up phone calls.
  Arms: Intervention group
Behavioral: Usual care — routine care including written mouth exercise instructions
  Arms: Control group

SUMMARY:
PURPOSE: The purpose of the study was to investigate the efficacy of mouth-opening training with follow-up on 1st、3rd、6th months for reducing postoperative trismus in patients with oral cancer.

METHODS: The study is a quasi-experimental design using repeated measures. 44 patients admitted at a general hospital in Taiwan for oral cancer surgery were recruited to the control group first then 38 patients were recruited to the intervention group. All subjects were instructed to practice mouth-opening exercises three times a day every day for three months and two telephone calls fellow up. Subjects in the intervention group received mouth-opening exercise adherence. Data on maximum interincisal opening and mandibular function impairment were collected before surgery, at one month, three months, and six months after radiotherapy, using the TheraBite Range-of-Motion scale and Mandibular Function Impairment Questionnaire, Restriction of Mouth Opening Questionnaire, and Difficulty of Food Intake.

DETAILED DESCRIPTION:
The purpose of the study was to investigate the effect of mouth-opening exercise training with follow-up telephone calls for preventing postoperative trismus in patients with oral cancer. The specific aims were to test the intervention effects on enhancing mouth-opening exercise practice, MIO, and mandibular function. We hypothesized that the intervention group would show 1) better adherence to mouth-opening exercises, 2) greater MIO, and 3) better mandibular function over time, compared to the control group.

The study is a quasi-experimental design with repeated measures. A convenience sample of 44 oral cancer patients was recruited to control group the 38 patients was recruited to the intervention group Subjects in the control group received routine care including written mouth exercise instructions. Subjects in both groups received two 30-minute individual trainings on the mouth-opening exercises before discharge from the hospital. Patients in the experimental group were provided with two one-on-one oral exercise instruction courses after receiving the last two radiation treatments by nurse practitioner. Subjects in the intervention group received additional 2 follow-up phone calls from the interventionist to enhance mouth-opening exercise adherence. Data on MIO and mandibular function impairment were collected before surgery, at one-month, three-months and six month after radiotherapy, using the TheraBite Range-of-Motion scale and the Mandibular Function Impairment Questionnaire. The study was approved by the research ethics committee of the hospital where the data were collected.

All statistical analyses were carried out using the SPSS statistical package version 20.0 (SPSS Inc., Chicago, IL, USA). Characteristics of the subjects were summarized by percentages, means, and standard deviations (SDs). Chi-squared tests or Fisher's exact tests and two independent samples t-tests were used to examine group baseline equivalency. Value changes of study outcomes (MIO and mandibular function impairment) and mouth-opening exercises performed from T1, T2, to T3 were expressed in two study groups. A general linear model was used to model these outcomes as a function of main group effect and main time effect. An interaction term (group difference by time) was added into each model to investigate the synergistic effect of the intervention with time. Both the stability analysis and the analysis of repeated relationships were performed by generalized estimation equations (GEE).

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. have a clear consciousness
3. can communicate in Mandarin and Taiwanese
4. diagnosed by a doctor as primary oral cancer (including gums, the floor of the mouth, buccal mucosa, hard palate, and posterior molar area) and
5. undergoing oral cancer tumor resection (including upper lymphatic removal) Those who have undergone skin flap reconstruction
6. radiation and/or concurrent chemotherapy.

Exclusion Criteria:

1. Poor wound healing after surgery and unable to perform the oral movement
2. no incisor or the position of the incisor after surgery is replaced by a flap due to surgery, the maximum opening distance cannot be measured
3. those with lip and tongue cancers that are less related to the closure of the teeth ( Or those who are physically unable to exercise)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-07-07 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2014-12-12 (Actual)

PRIMARY OUTCOMES:
MIO( Maximum inter-incisal opening) | Change from pre-intervention and during the intervention on 2, 4, and 6 months
  With the disposable oral activity scale (The TheraBite Range-of-Motion Scales), patients are asked to open their mouths as wide as possible while sitting on a chair. The TheraBite Range-of-Motion Scale was used to measure MIO with the subject in an upright position. Subjects with MIO <35 mm were considered to have trismus. The scale was measured by mm. For all values of mouth opening from 20 to 50 mm.The higher the score, the mouth is open.

SECONDARY OUTCOMES:
Restriction of Mouth Opening Questionnaire | Change from pre-intervention and during the intervention on 2, 4, and 6 months
  There are 10 questions in the questionnaire. The content includes the restriction on eating, speaking, cleaning, and inspection of the oral cavity. Each question is scored on a Likert scale with a score of 1-5. The average score of each question is the total score of the scale. The higher the score, the mouth is open. The higher the degree of restriction. Chinese translation version of the questionnaire, the expert validity of each question content validity index score is greater than 0.8, for oral cancer patients (n = 60) Cronbach's α is 0.96
Mandibular Function Impairment Questionnaire | Change from pre-intervention and during the intervention on 2, 4, and 6 months
  There are 17 questions, including the difficulty of chewing hard and soft foods, taking a big bite of food, laughing, eating specific foods, social activities, speaking, etc. Each question is scored on the Likert scale of 0-4 points. The scores of each question are added and divided by 68 to convert to a total score of 0-1 points. The higher the score, the more severe the functional impairment.
Exercise Time | each week during the intervention
  oral exercise practicing time recoded by participants by time of exercise. Time is calculated in minutes

CONTACTS AND LOCATIONS:
Overall Officials: SuFan Wu, Doctor, Study Director — National Taipei University of Nursing and Health Sciences

IPD SHARING:
Plan to Share IPD: No